CLINICAL TRIAL: NCT02798458
Title: Evaluation of the Gastrointestinal Manifestation of Fabry's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Braden Kuo, Instructor in Medicine, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015P000097
Record Dates: First submitted 2016-06-03; First posted 2016-06-14 (Estimated); Results first posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-02

CONDITIONS: Fabry's Disease
Keywords: Fabry's Disease; Fabry
MeSH Terms: conditions — Fabry Disease | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SmartPill Test (Experimental): All subjects will be asked to complete a SmartPill test. The SmartPill capsule is pill-shaped and about an inch long and ½ inch wide, or about the size of a vitamin pill. The receiver unit is about the size of a paperback book. The receiver gets signals from the capsule and stores the signals on a computer chip. The capsule detects the level of acidity, temperature, and pressures in your stomach and intestines and sends the information by radio wave signals to the receiver.
  Interventions: Device: Smartpill
- Endoscopic Mucosal Resection (Experimental): An additional small group of subjects will also be asked to complete a Sigmoidoscopy (an exam used to evaluate the lower part of the large intestine) during which an Endoscopic Mucosal Resection (removal of a small amount of tissue from the outermost layer of gut wall) will be completed. In the Endoscopy Mucosal Resection (EMR) procedure we will use an instrument called an endoscope (a lighted, flexible tube) to take a tissue sample from the rectum. This is the same type of instrument used in a routine colonoscopy
  Interventions: Device: Smartpill; Procedure: Endoscopic Mucosal Resection

INTERVENTIONS:
Device: Smartpill — The SmartPill Test is approved by the U.S. Food and Drug Administration (FDA) to measure transit time in the GI tract. This procedure uses the SmartPill capsule, a receiver, and computer software.
Procedure: Endoscopic Mucosal Resection — a Sigmoidoscopy is an exam used to evaluate the lower part of the large intestine) during which an Endoscopic Mucosal Resection (removal of a small amount of tissue from the outermost layer of gut wall) will be completed.
  Arms: Endoscopic Mucosal Resection

SUMMARY:
Patients will undergo a SmartPill test to gain additional understanding of Fabry disease manifestation via motility abnormalities in order to improve symptom targeted therapy. An additional Endoscopic mucosal resection may be performed on further qualifying patients. Tissue analysis from this biopsy will include evaluation of abnormalities of cellular structure and morphology with correlation with gastrointestinal complaints for each patient and comparison against age matched non-Fabry patient tissue. The hypothesis is that patients with fabry disease will have abnormal motility which will correlate with the patients symptoms and quality of life as noted on the questionnaires.

DETAILED DESCRIPTION:
Background: Gastrointestinal manifestations such as abdominal pain, diarrhea and nausea are prominent and, although typically non life-threatening, can frequently cause significant morbidity and burden in a patient with Fabry disease. Additional in depth understanding of gastrointestinal symptoms pathophysiology in Fabry disease is acutely needed in order to develop more specific evaluation of the symptoms and advance the treatment of these patients.

Hypothesis: Patients with gastrointestinal (GI) symptoms will have delayed motility on the SmartPill study, abnormal histologic findings on mucosal resection and symptoms that correlate with abnormal histologic and SmartPill findings. By gaining additional insight into the characterization of symptoms and the relationship to dysmotility, we anticipate improved and more focused adjunct therapies for the patients.

Methods: This study will consist of a screening visit, a SmartPill testing procedure visit, and a follow up visit for all subjects enrolled in the study. Fifteen of these patients, who clinically warranted sigmoidoscopy, will be asked to also complete an endoscopic mucosal resection (EMR) visit in addition to the other aspects of the study. Thus, each subject will report to the study site for at least 3 visits and up to 4 visits.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-70 years who have diagnosed Fabry disease either by enzyme testing in males or by enzyme and/or genetically confirmed mutation in females.
* Adults with Fabry disease having any gastrointestinal complaints within the past year.
* Endoscopic Mucosal Resection ONLY - Symptomatic subjects necessitating a sigmoidoscopy who are enzyme replacement therapy (ERT) naive OR less than 6 months of treatment.

Exclusion Criteria:

1. Fabry disease with other concomitant gastrointestinal diagnosis (Example:

   Inflammatory Bowel Disease, Celiac Disease)
2. Pregnancy
3. Endoscopic mucosal resection exclusions:

   1. Any contraindication to conscious sedation,
   2. Contraindication to endoscopy,
   3. Untreated or unmanageable coagulopathy,
   4. Thrombocytopenia (<50).
   5. Patient on ERT for more than 6 months.
4. Exclusions for SmartPill:

   1. Previous history of bezoars.
   2. Prior GI surgery except for cholecystectomy, appendectomy, or Nissen fundoplication.
   3. Any abdominal surgery within the past 3 months
   4. History of diverticulitis, diverticular stricture, and other intestinal strictures
   5. Tobacco use within eight hours prior to capsule ingestion and during the initial 8-hour recording on Day 0 or the Ingestion visit.
   6. Alcohol use within eight hours prior to capsule ingestion and throughout the entire monitoring period (5 days).
   7. BMI > 38
   8. Allergies to components of the SmartBar
   9. Use of medical devices such as pacemakers, infusion pumps, or insulin pumps.
   10. Uncontrolled diabetes with a hemoglobin A1C greater than 10.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-05; Primary Completion 2021-11-10 (Actual); Study Completion 2022-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Braden Kuo, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Bar N, Karaa A, Kiser K, Kuo B, Zar-Kessler C. Gastrointestinal Sensory Neuropathy and Dysmotility in Fabry Disease: Presentations and Effect on Patient's Quality of Life. Clin Transl Gastroenterol. 2023 Dec 1;14(12):e00633. doi: 10.14309/ctg.0000000000000633. PMID 37578052

RESULTS

PARTICIPANT FLOW:
Groups:
- SmartPill Test Only: All subjects will be asked to complete a SmartPill test. The SmartPill capsule is pill-shaped and about an inch long and ½ inch wide, or about the size of a vitamin pill. The receiver unit is about the size of a paperback book. The receiver gets signals from the capsule and stores the signals on a computer chip. The capsule detects the level of acidity, temperature, and pressures in your stomach and intestines and sends the information by radio wave signals to the receiver.
  Smartpill: The SmartPill Test is approved by the U.S. Food and Drug Administration (FDA) to measure transit time in the GI tract. This procedure uses the SmartPill capsule, a receiver, and computer software.
- SmartPill and Endoscopic Mucosal Resection: An additional small group of subjects will also be asked to complete a Sigmoidoscopy (an exam used to evaluate the lower part of the large intestine) during which an Endoscopic Mucosal Resection (removal of a small amount of tissue from the outermost layer of gut wall) will be completed. In the Endoscopy Mucosal Resection (EMR) procedure we will use an instrument called an endoscope (a lighted, flexible tube) to take a tissue sample from the rectum. This is the same type of instrument used in a routine colonoscopy
  Smartpill: The SmartPill Test is approved by the U.S. Food and Drug Administration (FDA) to measure transit time in the GI tract. This procedure uses the SmartPill capsule, a receiver, and computer software.
  Endoscopic Mucosal Resection: a Sigmoidoscopy is an exam used to evaluate the lower part of the large intestine) during which an Endoscopic Mucosal Resection (removal of a small amount of tissue from the outermost layer of gut wall) will be completed.
Period: Smart Pill Test (1 Day)
Arm/Group | SmartPill Test Only | SmartPill and Endoscopic Mucosal Resection
Started (48 patients total enrolled, 35 started and completed the SmartPill only and 13 started and completed the EMR and SmartPill.) | 35 | 13 (48 patients total enrolled, 35 started and completed the SmartPill only and 13 started and completed the EMR and SmartPill.)
Completed (48 patients total enrolled, 35 started and completed the SmartPill only and 13 started and completed the EMR and SmartPill.) | 35 | 13 (48 patients total enrolled, 35 started and completed the SmartPill only and 13 started and completed the EMR and SmartPill.)
Not Completed | 0 | 0
Period: Endoscopic Mucosal Resection (1 Day)
Arm/Group | SmartPill Test Only | SmartPill and Endoscopic Mucosal Resection
Started | 0 | 13
Completed | 0 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Reported demographics are separated by sex/gender.
Groups:
- Female; Male: Demographics
- Total: Total of all reporting groups
Arm/Group | Female | Male | Total
Number analyzed (Participants) | 28 | 20 | 48
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Self-Questionnaires
  years | 46 [32 to 57] | 46.5 [29 to 55] | 46.5 [32 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 0 | 28
  Male | 0 | 20 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 26 | 17 | 43
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 16 | 43
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 20 | 48
Enzyme replacement therapy > 6 months [Count of Participants; unit: Participants] | 15 | 13 | 28
Any neurologic involvement [Count of Participants; unit: Participants] | 27 | 19 | 46
Peripheral nervous system involvement [Count of Participants; unit: Participants] | 27 | 19 | 46
Central nervous system (serious) involvement - make clear this excludes CN [Count of Participants; unit: Participants] | 7 | 3 | 10
Cardiac system involvement [Count of Participants; unit: Participants] | 20 | 17 | 37
Renal systemic involvement [Count of Participants; unit: Participants] | 8 | 13 | 21
Dermatology systemic involvement [Count of Participants; unit: Participants] | 8 | 13 | 21
Ophthalmic systemic involvement [Count of Participants; unit: Participants] | 22 | 9 | 31
Psychiatric systemic involvement [Count of Participants; unit: Participants] | 20 | 6 | 26
Asthma systemic involvement [Count of Participants; unit: Participants] | 8 | 5 | 13
Presenting age of any neurologic systemic involvement [Median (Inter-Quartile Range); unit: years] | 7 [0 to 23] | 10 [1.3 to 16.8] | 9 [0 to 18]
Presenting age of cardiac systemic involvement [Median (Inter-Quartile Range); unit: years] | 34 [18 to 48] | 32 [22 to 40] | 32.5 [20.3 to 45]
Presenting age of renal systemic involvement [Median (Inter-Quartile Range); unit: years] | 20.5 [0 to 29.5] | 32 [16 to 52] | 28 [13.5 to 40]
Presenting age of ophthalmic systemic involvement [Median (Inter-Quartile Range); unit: years] | 15.5 [0 to 38] | 31 [13 to 40] | 24.5 [5.3 to 38]
Presenting age of psychiatric systemic involvement [Median (Inter-Quartile Range); unit: years] | 33.5 [21 to 45.3] | 36.5 [16.5 to 42.3] | 34.5 [23.8 to 43.3]
Presenting age of respiratory (asthma) systemic involvement [Median (Inter-Quartile Range); unit: years] | 20 [13.3 to 53.3] | 9 [5.5 to 32] | 19 [8 to 43]

OUTCOME MEASURES:

1. Primary Outcome: Gastric Emptying Transit Time Measured Via SmartPill Study
Description: The primary outcome of dysmotility will be the measurement of gastric emptying transit time via a SmartPill study. Delayed GET are defined as longer than 5 hours.
Time Frame: Up to 5 hours
Population: Demographics
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Female | Male
Number analyzed (Participants) | 28 | 20
Hours | 2.9 [2.5 to 3.8] | 2.8 [2.2 to 3.6]

2. Primary Outcome: Small Bowel Transit Time Measured Via SmartPill Study
Description: The primary outcome of dysmotility will be the measurement of small bowel transit time via a SmartPill study. Delayed SBTT are defined as longer than 6 hours.
Time Frame: Up to 6 hours
Population: Demographics
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Female | Male
Number analyzed (Participants) | 27 | 20
Hours | 4.3 [3.8 to 5] | 4.5 [3.1 to 5.6]

3. Primary Outcome: Colonic Transit Time Measured Via SmartPill Study
Description: The primary outcome of dysmotility will be the measurement of colonic transit time via a SmartPill study. Delayed CTT is defined as longer than 59 hours.
Time Frame: Up to 67 hours
Population: Demographics
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Female | Male
Number analyzed (Participants) | 27 | 20
Hours | 38.1 [20.3 to 66.8] | 21.3 [14.2 to 43.4]

4. Secondary Outcome: Gastrointestinal Symptom Assessment and Quality of Life, Work, and Productivity Via Questionnaires
Description: Participants will complete several questionnaires during study participation regarding gastrointestinal symptoms (lower and upper GI). These results will be used to determine overall gastrointestinal involvement and will be correlated with transit time and histologic findings
Time Frame: Up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Female | Male
Number analyzed (Participants) | 28 | 20
Participants
  Dysregulated bowel habits | 25 | 17
  Reporting chronic diarrhea | 14 | 16
  Reporting chronic constipation | 20 | 11
  Reporting only diarrhea | 5 | 6
  Reporting only constipation | 11 | 1
  Chronic abdominal pain | 25 | 14
  Symptoms compatible with IBS | 23 | 14
  Bloating | 23 | 10
  Functional dyspepsia | 26 | 13
  Dysphagia | 2 | 0
  nausea and vomiting | 15 | 7
  Gastroesophageal reflux disease symptoms | 15 | 2
  Moderate severe depression | 4 | 0
  Moderate severe anxiety | 18 | 13
  Unemployed by Work Productivity and Activity Impairment | 5 | 9
  Work loss- 40% and more by Work Productivity and Activity Impairment | 2 | 2
  Reduced productivity 40% and more by Work Productivity and Activity Impairment | 9 | 3
  Work/productivity impairment by Work Productivity and Activity Impairment | 14 | 13

5. Secondary Outcome: Age of Symptom Start
Time Frame: Up to 4 weeks
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | Female | Male
Number analyzed (Participants) | 28 | 20
years
  Age of first gastrointestinal symptoms | 15 [0.5 to 26.5] | 10 [6.8 to 18]
  Age of abdominal pain symptom start | 25 [10 to 39.5] | 10 [9.5 to 16]
  Age of Diarrhea symptom start | 16 [7 to 40] | 10 [0 to 12]
  Age of constipation symptom start | 15 [8 to 27.5] | 15 [3 to 42.8]
  Age of nausea symptom start | 28 [15 to 49] | 20 [19 to 25]
  Age of vomiting symptom start | 13 [13 to 13] | 20 [20 to 20]

6. Secondary Outcome: Delayed Gastric Emptying Measured Via SmartPill Study
Description: The secondary outcome of dysmotility will be the measurement of delayed gastric emptying measured via a SmartPill study. Delayed GET are defined as longer than 5 hours.
Time Frame: Up to 5 hours
Population: Demographics
Measure: Count of Participants; unit: Participants
Arm/Group | Female | Male
Number analyzed (Participants) | 27 | 20
Participants | 3 | 2

7. Secondary Outcome: Delayed Small Bowel Transit Measured Via SmartPill Study
Description: The secondary outcome of dysmotility will be the measurement of delayed bowel transit time via a SmartPill study. Delayed SBTT are defined as longer than 6 hours.
Time Frame: Up to 6 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Female | Male
Number analyzed (Participants) | 27 | 20
Participants | 1 | 2

8. Secondary Outcome: Delayed Colonic Transit Measured Via SmartPill Study
Description: The secondary outcome of dysmotility will be the measurement of delayed colonic transit time via a SmartPill study. Delayed CTT is defined as longer than 59 hours.
Time Frame: Up to 67 hours
Population: Demographics
Measure: Count of Participants; unit: Participants
Arm/Group | Female | Male
Number analyzed (Participants) | 27 | 20
Participants | 8 | 2

9. Secondary Outcome: Symptom Severity Index
Description: Patient reported severity of certain symptoms over the last 4 weeks on a scale of 0 to 10 (bloating, abdominal discomfort, incomplete evacuation, straining and urgency). Higher score would mean worse (more symptoms) outcome.
Time Frame: At 67 hours, data reported over the last 4 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Female | Male
Number analyzed (Participants) | 28 | 20
score on a scale
  Bloating | 6 [2.3 to 8] | 2 [0 to 4.5]
  Abdominal discomfort | 6.5 [3 to 7] | 4 [2 to 6]
  Sense of incomplete evacuation | 3.5 [2 to 7] | 2 [0 to 4]
  Straining while defecating | 3.5 [2 to 6.8] | 1.5 [0 to 4]
  Bowel urgency | 4 [2.3 to 7.8] | 4 [2 to 6.8]

10. Secondary Outcome: Symptom Frequency Assessment (SFA)
Description: Patients reported the number of complete BMs they had during the last week (minimum could be 0 and the maximum could be any number greater than 0). Higher/lower scores could be the better or worse outcome (e.g., 0 bowel movements all week would be a worse outcome but over 10 bowel movements would be worse as well), it just depends on the extent.
Time Frame: At 67 hours, data reported over the last 7 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Female | Male
Number analyzed (Participants) | 28 | 20
units on a scale
  Daily bowel movements | 1 [1 to 2] | 2.5 [1 to 4]
  Weekly bowel movements | 5.5 [3.6 to 13.5] | 16 [10 to 25]

11. Secondary Outcome: Hamilton Anxiety Rating Scale (HAM-A)
Description: The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <7 indicates no or minimal severity, 8-14 is mild anxiety, 15-23 is moderate anxiety and 24 and worse is severe anxiety 5. Moderate-severe anxiety was defined as a score of 15 and above.
Time Frame: At 4 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Female | Male
Number analyzed (Participants) | 28 | 20
score on a scale | 16.5 [12 to 20] | 16.5 [4 to 18.8]

12. Secondary Outcome: Beck's Depression Inventory (BDI)
Description: Beck's Depression Inventory (BDI): is a 21-item tool assessing the existence and severity of symptoms of depression, as defined by the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV; 1994). The items correspond to symptoms of depression and are a four-point scale for each item ranging from 0 to 3. They are summed to give a single BDI score between 0-63 (where higher results reflect more severe depression). Grades are 1-10: normal, 11-16: mild mood disturbance, 17-20: borderline clinical depression, 21-30: moderate depression, 31-40: severe depression, and >40 extreme depression 6. Moderate-severe depression was defined as a score of 21 and above.
Time Frame: At 4 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Female | Male
Number analyzed (Participants) | 28 | 20
score on a scale | 10.5 [6 to 14.8] | 6.5 [2.3 to 14]

13. Secondary Outcome: Work Productivity and Activity Impairment (WPAI)
Description: Work Productivity and Activity Impairment (WPAI): examines the effect of GI symptoms on loss of work time and loss of productivity. Patients indicated if they are unemployed. For employed patients, scores are presented as percentage of time lost during the last week (hours lost due to GI symptoms out of the hours that patient should have worked, excluding the time lost on participating in the study). Higher percentages indicate greater impairment. Work missed percentage, reduced productivity percentage, and work-productivity impairment percentage (combining the 2 scores) are calculated 7. We defined work/productivity impairment as either being unemployed or having lost 40% or more of work time or productivity. For employed patients, scores are presented as percentage of time lost during the last week (hours lost due to GI symptoms out of the hours that patient should have worked, excluding the time lost on participating in the study).
Time Frame: At 7 days
Measure: Median (Inter-Quartile Range); unit: percentage of time lost during the last
Arm/Group | Female | Male
Number analyzed (Participants) | 28 | 20
percentage of time lost during the last
  work missed (%) | 0 [0 to 0] | 0 [0 to 10.8]
  reduced productivity while working (%) | 20 [10 to 50] | 10 [10 to 50]
  work productivity impairment (%) | 20 [10 to 52.1] | 10 [10 to 60]

14. Secondary Outcome: IBS Quality of Life (IBS QoL) and Sub-scores
Description: Irritable bowel syndrome quality of life (IBS-QOL): Assesses bowel specific QOL. It consists of 34 items of a 5-point Likert scale. The total score is summed and then transformed to a 0-100 scale, where 0 is low QoL, and 100 is the best QoL. Different IBS-QOL items can also be categorized to eight subscale scores (Dysphoria, Interference with Activity, Body Image, Health Worry, Food Avoidance, Social Reaction, Sexual, Relationships). Note be made, that the IBS-QOL examines the effect of "bowel problems" on different aspect of QOL, and so was used to assess the effect of gut symptoms on the patients' QOL. Higher scores are better outcome.
Time Frame: At 4 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Female | Male
Number analyzed (Participants) | 28 | 20
score on a scale
  Dysphoria sub-score | 85.7 [70 to 95.7] | 85.7 [59.3 to 93.6]
  Interference with Activity sub-score | 57.1 [39.3 to 71.4] | 46.4 [30.4 to 60.7]
  Body Image sub-score | 68.8 [53.1 to 81.3] | 87.5 [75 to 100]
  Health Worry sub-score | 75 [62.5 to 91.7] | 83.3 [77.1 to 91.7]
  Food avoidance sub-score | 50 [33.3 to 87.5] | 75 [43.8 to 89.6]
  Social reaction sub-score | 87.5 [71.9 to 96.9] | 84.4 [68.8 to 98.4]
  Sexual sub-score | 100 [68.8 to 100] | 100 [78.1 to 100]
  Relationships sub-score | 100 [79.2 to 100] | 91.7 [77.1 to 100]
  IBS-QOL | 80.2 [61.8 to 89] | 81.6 [65.1 to 87.9]

15. Secondary Outcome: Bristol Stool Scale
Description: Bristol Stool Scale: patients indicate their last 7 days stool consistency on 1-7 visual scale. The Bristol stool scale correlates with colonic transit time. Higher scores do not indicate better or worse outcomes. It is a visual scale.
Time Frame: At 7 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Female | Male
Number analyzed (Participants) | 28 | 20
score on a scale | 4 [2 to 5] | 6 [4 to 6]

ADVERSE EVENTS:
Time Frame: Up to 4 days
Arm/Group | SmartPill Test | Endoscopic Mucosal Resection
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/13
Other Adverse Events (participants affected / at risk) | 1/48 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SmartPill Test (N=48) | Endoscopic Mucosal Resection (N=13)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) — 06/27/2017
syncope (Gastrointestinal disorders) | 1 (1) | 1 (1) — 06/27/2017
ER visit (Gastrointestinal disorders) | 1 (1) | 1 (1) — 06/27/2017
Fever (Gastrointestinal disorders) | 1 (1) | 1 (1) — 07/17/2019
Rectal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) — 07/16/2019

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT02798458/Prot_SAP_000.pdf